CLINICAL TRIAL: NCT05361772
Title: Low-dose Colchicine Inhibit Abdominal Aortic Aneurysm Growth Trial
Acronym: COIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Shenzhen People's Hospital (Other); Peking University Shougang Hospital (Other); Peking Union Medical College Hospital (Other); Second Xiangya Hospital of Central South University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Shenzhen Bao an People's Hospital (Unknown)
Responsible Party: Principal Investigator, Jianfang Luo, chief physician, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY-N-2022-027-03
Record Dates: First submitted 2022-04-30; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Colchicine; Abdominal Aortic Aneurysm; Progression
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Disease Progression | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose colchicine group (Experimental): colchicine 0.5mg per day for 24 months
  Interventions: Drug: colchicine
- placebo group (Placebo Comparator): placebo 0.5mg per day for 24 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: colchicine — colchicine 0.5mg per day for 24 months
  Arms: low-dose colchicine group
Drug: Placebo — placebo 0.5mg per day for 24 months
  Arms: placebo group

SUMMARY:
COIN trial is a a prospective, randomized, placebo-controlled, double-blind, multicenter clinical study. Approximately 230 patients with small abdominal aortic aneurysms (AAA) will be randomly allocated to low-dose colchicine group or placebo group. All study patients will be followed up in the outpatient clinic every 3 months and undergo CTA scans after 24 months from randomization. The primary objective is to test the hypothesis that low dose colchicine can inhibit the progression of AAA diameter. The secondary objective is to test the hypothesis that low dose colchicine can inhibit the progression of AAA volume, reduce the incidence of clinical outcomes associated with AAA, reduce the incidence of major adverse cardiovascular events and all-cause mortality.

DETAILED DESCRIPTION:
This study is a prospective, randomized, placebo-controlled, double-blind, multicenter clinical study to test the research hypothesis that low-dose colchicine (0.5 mg/d) can delay the progression of AAA.

The study will enroll patients with infrarenal abdominal aortic aneurysms with a maximum diameter of 30-50 mm and no indication for surgical or endovascular treatment. All patients will receive the best standard medical treatment. Before randomization, all patients will undergo a 1-month lead-in period, during which open-label colchicine 0.5 mg/d will be administered. If there is colchicine intolerance, they will not be randomized.

The study center performed computer-generated block randomization (block size 8). Randomization method and block size will not unblinded until all data analyses are completed. Enrolled patients will randomly assigned to each hospital in a 1:1 ratio by the randomization center through sequentially coded, sealed, light-tight envelopes, to colchicine and placebo groups.

After randomization, patients will receive low-dose colchicine (0.5 mg/d) or placebo, respectively, and will be followed up for 24 months. We will evulate whether low-dose colchicine can delay the progression of AAA by assessing the change in maximum aneurysm diameter by CTA. At the same time, its effects on abdominal aortic aneurysm-related and cardiovascular-related clinical events will be observed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged over 55 and under 85; 2. Diagnosis of infrarenal abdominal aortic aneurysm within 3 months by CTA; 3. No indication for endovascular repair or surgery of abdominal aortic aneurysm

Exclusion Criteria:

* 1. Currently using colchicine; 2. Allergic to colchicine; 3. History of abdominal aortic aneurysm repair or surgery; 4. Combined with aortic dissection, thoracic aortic aneurysm, penetrating aortic ulcer (ulcer width>2cm and depth>1cm) and other aortic diseases requiring intervention; 5. Abdominal aortic aneurysm involving the renal artery or suprarenal abdominal aortic aneurysm; 6.Diameter of iliac aneurysm >29mm; 7. Renal artery stenosis or iliac artery stenosis planned for immediate intervention; 8. AAA caused by connective tissue disease (eg, collagen vascular disease), hereditary or genetic syndrome (eg, Marfan syndrome, Ehlers-Danlos syndrome); 9. Severe renal dysfunction (serum creatinine >176.8umol/L or eGFR <30ml/min) in the last 3 months 10. Severe liver dysfunction (ALT>2 ULN or TBIL>2 ULN)in the last 3 months; 11.Abnormal blood routine (hemoglobin <115g/L, white blood cell count<3.0×10^9/L, or platelet count <110×10^9/L) in the last 3 months; 12. Presence of inflammatory bowel disease or chronic diarrhea; 13. Current or planned usage of systemic immunosuppressants (eg, prednisone, azathioprine, methotrexate, cyclosporine for autoimmune disease or after bone marrow, heart, liver, lung, or other solid organ transplantation) ; 14.Patients with malignant tumors and autoimmune diseases; 15. Unable to take care of themselves, frail or expected survival time < 2 years; 16. Peripheral neuritis, myositis, or statin-related elevation of muscle enzymes; 17. Premenopausal, pregnant or lactating female patients; 18. Participated in other clinical studies of interventional therapy or drug therapy, which may interfere with the research results; 19. Refused or unable to sign informed consent to enter clinical research or to follow the research protocol and follow up.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of the maximum diameter of abdominal aortic aneurysm | 24 months
  the changes of the maximum diameter of abdominal aortic aneurysm on CTA in 24 months

SECONDARY OUTCOMES:
changes of the maximum volume of abdominal aortic aneurysm | 24 months
  the changes of the maximum volume of abdominal aortic aneurysm on CTA in 24 months
aorta-related adverse events | 24 months
  rupture of abdominal aortic aneurysm, endovascular repair or surgery repair of abdominal aortic aneurysm,aortic-related death
major adverse cardiovascular events | 24 months
  cardiovascular death, acute coronary syndrome, interventon for coronary artery disease, ischemic stroke or transient ischemic attack
all-cause mortality | 24 months
  all-cause mortality
aortic-related mortality | 24 months
  aortic-related mortality
cardiovascular -related mortality | 24 months
  cardiovascular -related mortality
change of inflammatory biomarkers | 24 months
  change of CRP，D-dimer，MMP-9, IL-1β, IL-18
change of living quality | 24 months
  SF - 36 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jianfang Luo, MD, Study Chair — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sakalihasan N, Michel JB, Katsargyris A, Kuivaniemi H, Defraigne JO, Nchimi A, Powell JT, Yoshimura K, Hultgren R. Abdominal aortic aneurysms. Nat Rev Dis Primers. 2018 Oct 18;4(1):34. doi: 10.1038/s41572-018-0030-7. PMID 30337540
- [Background] Li W, Luo S, Luo J, Liu Y, Ning B, Huang W, Xue L, Chen J. Predictors Associated With Increased Prevalence of Abdominal Aortic Aneurysm in Chinese Patients with Atherosclerotic Risk Factors. Eur J Vasc Endovasc Surg. 2017 Jul;54(1):43-49. doi: 10.1016/j.ejvs.2017.04.004. Epub 2017 May 17. PMID 28527818
- [Background] Guirguis-Blake JM, Beil TL, Senger CA, Coppola EL. Primary Care Screening for Abdominal Aortic Aneurysm: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2019 Dec 10;322(22):2219-2238. doi: 10.1001/jama.2019.17021. PMID 31821436
- [Background] Kuivaniemi H, Elmore JR. Opportunities in abdominal aortic aneurysm research: epidemiology, genetics, and pathophysiology. Ann Vasc Surg. 2012 Aug;26(6):862-70. doi: 10.1016/j.avsg.2012.02.005. PMID 22794334
- [Background] Umebayashi R, Uchida HA, Wada J. Abdominal aortic aneurysm in aged population. Aging (Albany NY). 2018 Dec 6;10(12):3650-3651. doi: 10.18632/aging.101702. No abstract available. PMID 30523221
- [Background] Liu CL, Ren J, Wang Y, Zhang X, Sukhova GK, Liao M, Santos M, Luo S, Yang D, Xia M, Inouye K, Hotamisligil GS, Lu G, Upchurch GR, Libby P, Guo J, Zhang J, Shi GP. Adipocytes promote interleukin-18 binding to its receptors during abdominal aortic aneurysm formation in mice. Eur Heart J. 2020 Jul 7;41(26):2456-2468. doi: 10.1093/eurheartj/ehz856. PMID 31821481
- [Background] Golledge J. Abdominal aortic aneurysm: update on pathogenesis and medical treatments. Nat Rev Cardiol. 2019 Apr;16(4):225-242. doi: 10.1038/s41569-018-0114-9. PMID 30443031
- [Background] Oliver-Williams C, Sweeting MJ, Jacomelli J, Summers L, Stevenson A, Lees T, Earnshaw JJ. Safety of Men With Small and Medium Abdominal Aortic Aneurysms Under Surveillance in the NAAASP. Circulation. 2019 Mar 12;139(11):1371-1380. doi: 10.1161/CIRCULATIONAHA.118.036966. PMID 30636430
- [Background] Freiberg MS, Arnold AM, Newman AB, Edwards MS, Kraemer KL, Kuller LH. Abdominal aortic aneurysms, increasing infrarenal aortic diameter, and risk of total mortality and incident cardiovascular disease events: 10-year follow-up data from the Cardiovascular Health Study. Circulation. 2008 Feb 26;117(8):1010-7. doi: 10.1161/CIRCULATIONAHA.107.720219. Epub 2008 Feb 11. PMID 18268154
- [Background] Forsythe RO, Dweck MR, McBride OMB, Vesey AT, Semple SI, Shah ASV, Adamson PD, Wallace WA, Kaczynski J, Ho W, van Beek EJR, Gray CD, Fletcher A, Lucatelli C, Marin A, Burns P, Tambyraja A, Chalmers RTA, Weir G, Mitchard N, Tavares A, Robson JMJ, Newby DE. 18F-Sodium Fluoride Uptake in Abdominal Aortic Aneurysms: The SoFIA3 Study. J Am Coll Cardiol. 2018 Feb 6;71(5):513-523. doi: 10.1016/j.jacc.2017.11.053. PMID 29406857
- [Background] MA3RS Study Investigators. Aortic Wall Inflammation Predicts Abdominal Aortic Aneurysm Expansion, Rupture, and Need for Surgical Repair. Circulation. 2017 Aug 29;136(9):787-797. doi: 10.1161/CIRCULATIONAHA.117.028433. Epub 2017 Jul 18. PMID 28720724
- [Background] Vainas T, Lubbers T, Stassen FR, Herngreen SB, van Dieijen-Visser MP, Bruggeman CA, Kitslaar PJ, Schurink GW. Serum C-reactive protein level is associated with abdominal aortic aneurysm size and may be produced by aneurysmal tissue. Circulation. 2003 Mar 4;107(8):1103-5. doi: 10.1161/01.cir.0000059938.95404.92. PMID 12615785